CLINICAL TRIAL: NCT00819286
Title: A Prospective, Randomized-Controlled, Multicenter Study Evaluating Primary Plating in High-Risk Median Sternotomy Patients for Osteosynthesis and Pain
Brief Title: Evaluation of Primary Plating in Sternotomy Patients for Osteosynthesis and Pain
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07071
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Results first posted 2012-03-15 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Sternal Wound Infection; Sternal Non-union; Pain; Mediastinitis
Keywords: open heart surgery
MeSH Terms: conditions — Pain; Mediastinitis | interventions — Bone Wires

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant blinded to treatment assignment until completion of study.
Oversight: Data Monitoring Committee: No

ARMS (2):
- wire (control) (Active Comparator): patients will have their sternum closed using wire (stainless steel surgical wire).
  Interventions: Device: wire (control)
- SternaLock Rigid Fixation Plates (Experimental): patients will have their sternum closed by rigid fixation using SternaLock Rigid Fixation Plates.
  Interventions: Device: SternaLock Rigid Fixation Plates

INTERVENTIONS:
Device: SternaLock Rigid Fixation Plates — patients will have their sternum closed by rigid fixation using SternaLock Rigid Fixation Plates
  Arms: SternaLock Rigid Fixation Plates
Device: wire (control) — patients will have their sternum closed using wire (stainless steel surgical wire).
  Arms: wire (control)

SUMMARY:
The goal of this study is to evaluate sternal osteosynthesis, chest wall pain and return to normal activity in open heart surgery patients who had their breast bone closed either with wires or plates.

DETAILED DESCRIPTION:
Median sternotomy patients will be randomized to either wire or rigid fixation groups. A scheduled evaluation period will record clinical parameters. Enrollment has ended with one hundred forty (140) patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing median sternotomy;
* Patients eighteen (18) years of age or older;
* Patients presenting two or more risk factors such as diabetes mellitus, Chronic Obstructive Pulmonary Disease, obesity (BMI > 30), osteoporosis, Renal failure, Chronic steroid use, Immunosuppression, Redo sternotomy, Neurologic dysfunction severely affecting ambulation,
* Off mid-line sternotomy
* bilateral IMA use
* Long cardio-pulmonary bypass runs
* Transverse fractures of the sternum

Exclusion Criteria:

* Patients with a non-standard sternotomy;
* Patients with an off-midline sternotomy that reduced the bony margin to <2mm
* Patients under eighteen (18) years of age;
* Patients that are pregnant or currently lactating;
* Patients presenting intra-operative conditions that would require the use of rigid fixation and/or additional post-sternotomy mechanical support beyond wire cerclage due to surgical evaluation,
* Patients defined within the New York Heart Association (NYHA) or Canadian Cardiovascular Society (CCS) functional Class IV for congestive heart failure,
* Patients presenting emergent/salvage cardiac acuity as defined per the Society of Thoracic Surgeons (STS) guidelines: i.e., patients undergoing cardiopulmonary resuscitation en route to the operating room or prior to induction of anesthesia;
* Patients undergoing post-operative revision procedures that treat the original sternotomy in such a way as to affect outcome (antibiotic irrigation, debridement or other treatment to the osteotomy);
* Patients unwilling or unable to return for follow-up;
* Lacking the ability to follow instructions;
* Intraoperative death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jai Raman, MD, Study Chair — University of Chicago; Michael Wong, MD, Principal Investigator — University of California Davis Medical Center, Sacramento, CA; Brian DeGuzmann, MD, Principal Investigator — St. Joseph's Medical Center, Phoenix, AZ; Sven Lehmann, MD, Principal Investigator — Leipzig Heart Center, Leipzig, Germany; Kenton Zehr, MD, Principal Investigator — Scott & White Memorial Hospital, Temple, TX; H Edward Garrett, Jr, MD, Principal Investigator — Baptist Memorial Hospital, Memphis, TN
Locations (6):
- United States (5):
  - St. Joseph's Heart and Lung Institute, Phoenix, Arizona
  - University of California Davis Medical Center, Sacramento, California
  - University of Chicago, Chicago, Illinois
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Scott & White Memorial Hospital, Temple, Texas
- Leipzig Heart Center, Leipzig, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective, randomized trial at 5 US sites and 1 European site. Patient enrollment occurred between November 2008 and May 2010.
Pre-assignment Details: Patients were randomized at the time of sternal closure to either rigid plate fixation or wire cerclage. A total of 140 patients were enrolled in this study (70 in each treatment group) and included in an intent to treat analysis.
Groups:
- Wire (Control): patients will have their sternum closed using stainless steel wires.
- Plates: patients will have their sternum closed by rigid fixation using SternaLock plates.
Period: Overall Study
Arm/Group | Wire (Control) | Plates
Started | 70 | 70
Completed | 56 | 45
Not Completed | 14 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wire (Control) | Plates | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (8.9) | 66.3 (9.8) | 65.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 52 | 51 | 103

OUTCOME MEASURES:

1. Primary Outcome: CT Scan Evaluation of Sternal Bone Healing
Description: Quantitative evaluation of sternal bone healing at 5 anatomical locations along the sternum using a 6 point quantitative scale (0= no healing and 5= complete healing)
Time Frame: 3 and 6 Months
Population: Patients were randomized to receive a CT scan at either 3 or 6 months. All patients who received a CT scan were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wire (Control) | Plates
Number analyzed (Participants) | 48 | 46
units on a scale
  3 Month CT Scan (n=25 wire, n=27 plates) | 0.9 (0.8) | 1.7 (1.1)
  6 Month CT Scan (n=26 wire, n=23 plates) | 2.2 (1.1) | 3.2 (1.6)
Statistical Analysis 1: Comparison: Wire (Control) vs Plates; 3 Month CT Scores (Plates vs Wires); Test type: Superiority or Other; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = 0
Statistical Analysis 2: Comparison: Wire (Control) vs Plates; 6 Month CT Scores (Plates vs Wires); Test type: Superiority or Other; p = 0.01, t-test, 2 sided

2. Primary Outcome: Activity Based Total Visual Analog Pain Score
Description: Postoperative VAS pain scores (scale of 0-10 for each; 0= no pain, 10= worst pain imaginable) were evaluated as a function of resting, coughing, sneezing and general movement. The sum of these was used to derive an "Activity Based Total Visual Analog Pain Score", (scale of 0-40; 0= no pain, 40= worst pain imaginable). For this primary endpoint analysis, the total score at 6 months was evaluated.
Time Frame: 6 months
Population: All patients with VAS pain data at 6 months were included in the analysis of the primary endpoint Activity Based Total Visual Analog Pain Score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wire (Control) | Plates
Number analyzed (Participants) | 56 | 44
units on a scale | 7.28 (4.65) | 7.20 (4.04)
Statistical Analysis 1: Comparison: Wire (Control) vs Plates; Plates vs Wires; Test type: Superiority or Other; p = 0.93, t-test, 1 sided; Mean Difference (Final Values) = 0

ADVERSE EVENTS:
Time Frame: 0 to 6 months
Description: Adverse events were classified for severity and causality
Arm/Group | Wire (Control) | Plates
Serious Adverse Events (participants affected / at risk) | 24/70 | 32/70
Other Adverse Events (participants affected / at risk) | 20/70 | 24/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wire (Control) (N=70) | Plates (N=70)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 3 (4)
Cardiac arrhythmias (Cardiac disorders) | 2 (2) | 2 (2)
Congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Low cardiac output (Cardiac disorders) | 2 (2) | 0 (0)
Multiple organ failure due to disecting aorta (Cardiac disorders) | 1 (1) | 0 (0)
Pacemaker implantation (Cardiac disorders) | 0 (0) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 0 (0) | 2 (2)
Convulsion (General disorders) | 1 (1) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Suspicion of lung fibrosis; bronchitis ongoing (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 2 (3) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2)
Resternotomy (Surgical and medical procedures) | 7 (7) | 11 (11)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wire (Control) (N=70) | Plates (N=70)
Cardiac arrhythmias (Cardiac disorders) | 9 (9) | 12 (12)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator may publish his/her own results from the study provided such publication does not include or disclose any confidential information. Principal investigator may also participate in joint publications. All proposed publications shall be submitted to Biomet for review. Biomet will have 30 days to review the proposed publication.